CLINICAL TRIAL: NCT07047690
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study of Nemolizumab in Adult Patients With Systemic Sclerosis
Brief Title: A Study of Nemolizumab for the Treatment of Adults With Systemic Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR207796
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-11

CONDITIONS: Systemic Sclerosis
Keywords: Limited Cutaneous Systemic Sclerosis; Diffuse Cutaneous Systemic Sclerosis; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Limited; Scleroderma, Diffuse; Lung Diseases, Interstitial | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nemolizumab Dose 1 (Experimental)
  Interventions: Drug: Nemolizumab
- Nemolizumab Dose 2 (Experimental)
  Interventions: Drug: Nemolizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab — Subcutaneous Injection
  Other Names: CD14152
  Arms: Nemolizumab Dose 1; Nemolizumab Dose 2
Drug: Placebo — Subcutaneous Injection
  Arms: Placebo

SUMMARY:
The main purpose of the study is to investigate the efficacy on cutaneous thickness and the safety of Nemolizumab in adult patients with systemic sclerosis after a 52-week treatment period and to select the optimal dose for this target population.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 18 years of age or older, at the time of signing the Informed Consent Form.
2. Classification of systemic sclerosis (SSc) as defined by the 2013 American College of Rheumatology [ACR]/European League Against Rheumatism [EULAR] criteria.
3. Modified Rodnan Skin Score.

   1. Diffuse cutaneous systemic sclerosis (DcSSc) participants and modified Rodnan Skin Score (mRSS) of greater than equal to (>=)12 and less than (<)30 at both screening and baseline
   2. Limited cutaneous systemic sclerosis (LcSSc) participants with mRSS >=8 at both screening and baseline. LcSSc participants with positive anti-centromere at screening are excluded.
4. Disease duration in DcSSc participants <= 5 years from screening and LcSSc participants <=2 years from screening is defined as the time from the first non-Raynaud's phenomenon manifestation of SSc.
5. Participants are permitted to receive the following background therapies stable for at least 3 months prior to baseline, including any combination of the following:

   1. Nintedanib (<150mg twice daily) and/or
   2. One of the following:

      1. Methotrexate (MTX) (<25mg weekly) or
      2. Mycophenolate mofetil (MMF), mycophenolate sodium (MPS), or mycophenolic acid (MPA) (<3000mg daily MMF, <2160mg daily for MPS or MPA) NOTE: MTX should not be used in combination with MMF/MPS/MPA
6. Participants with evidence for active or progressive disease.
7. Men (whose female partner can become pregnant) and women of childbearing potential will be required to use effective means of contraception or commit to true abstinence, when this is in line with preferred and usual lifestyle of the participant, during the study and for at least 12 weeks after receiving the last study treatment.
8. Female participants of non-childbearing potential
9. Signed informed consent

Exclusion Criteria:

1. Anti-centromere antibody positive at screening for participants with LcSSc.
2. Anti-RNA polymerase 3 antibody positive for participants with a disease duration >18months.
3. Creatinine clearance <30 milli liter per minute [ml/min] (calculated by Cockcroft-Gault formula).
4. Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HbcAb], hepatitis C [HCV] antibody with positive confirmatory test for hepatitis C virus [HCV] antibody with positive HCV RNA, or human immunodeficiency virus [HIV] antibody).
5. FVC <50% of predicted normal value, and DLCO <40% of predicted normal value (corrected for Hb) at screening and baseline.
6. Known diagnosis of clinically significant respiratory disorders other than ILD, including severe chronic obstructive pulmonary disease, severe asthma, recent (within 3 months) severe respiratory infections or history of recurrent respiratory infections, smoking, and any other respiratory condition that, in the opinion of the investigator, could interfere with the study or pose a risk to the participant.
7. Currently listed and/or anticipated to be listed for lung transplantation within the next 12 months.
8. Cardiovascular disease with clinically significant arrhythmia requiring therapy, congestive heart failure (New York Heart Association Class III-IV functional capacity), unstable angina, uncontrolled hypertension, Cor pulmonale, or symptomatic pericardial effusion.
9. History of myocardial infarction in the last 6 months prior to screening.
10. Pulmonary hypertension WHO Functional Class III or higher (as defined by WHO 2009) requiring treatment.
11. Clinical signs of severe malabsorption in the opinion of the investigator or needing parenteral nutrition.
12. History of scleroderma renal crisis (SRC) 6 months prior to screening.
13. Participants with underlying chronic liver disease (Child Pugh A, B, C hepatic impairment).
14. Body weight of <30.0 kilogram (Kg) at screening or BL
15. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed, or unwilling to use appropriate contraception measures during the study period
16. Previous treatment with nemolizumab
17. Participants with the primary diagnosis of a rheumatic autoimmune disease other than SSc, including but not limited to rheumatoid arthritis, systemic lupus erythematosus, polymyositis, dermatomyositis, systemic vasculitis, Sjogren's syndrome, anti-synthetase syndrome, or mixed CTD, as determined by the investigator with consultation of the medical monitors
18. Systemic sclerosis-like illness including but not limited to localized scleroderma (morphea), eosinophilic fasciitis, sclerodermoid graft-versus-host disease, fibro mucinous conditions (scleredema, scleromyxedema), scleroderma-like conditions that are associated with environmental chemical and drug exposure (e.g., toxic rapeseed oil, vinyl chloride, bleomycin, gadolinium-based contrast agents [nephrogenic systemic fibrosis], or due to metabolic disease)
19. History of hypersensitivity (including anaphylaxis) to an immunoglobulin product (plasma-derived or recombinant, e.g., monoclonal antibody) or to any of the study treatment excipient
20. Known active bacterial, viral, fungal, or any major episode of infection requiring hospitalization or treatment with IV antibiotics or antivirals within 4 weeks prior to screening, or oral antibiotics within 2 weeks prior to screening. Participants may be rescreened once the infection has resolved.
21. History of a primary immunodeficiency
22. History of Bone Morrow Transplantation. Chimeric Antigen Receptor (CAR)-T Cell Therapy or any other genetically engineering cells
23. History of lymphoproliferative disease or history of malignancy of any organ system within the last 5 years, except for (1) basal cell carcinoma, squamous cell carcinoma in situ (Bowen's disease), or carcinomas in situ of the cervix that have been treated and have no evidence of recurrence in the last 12 weeks before the BL visit, or (2) actinic keratoses that have been treated
24. History of alcohol or substance abuse dependence or any condition that, in the investigator's opinion makes the participant unreliable to following instructions and complete the study
25. In the opinion of the investigator, the participant has any medical condition, including clinically significant pulmonary abnormalities, or psychological condition,or clinically significant laboratory abnormalities that could pose undue risk to the participant, prevent study completion or adversely affect the validity or interpretability of the study measurements or interfere with the study assessments, or impede the participant's ability to complete the study.
26. Participant has not adhered to the restrictions in select treatments prior to screening or is not expected to be compliant with restrictions during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-05-28 (Estimated); Study Completion 2028-07-23 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline (BL) in Modified Rodnan Skin Score (mRSS) at Week 52 | Baseline, at Week 52
  mRSS is the assessment of skin involvement includes semiquantitative estimation of skin thickness, pliability (hardness), and fixation to underlying structures (tethering).Cutaneous thickness is assessed in 17 body surface areas using a 0-3 scale, where mRSS of score 0="normal" with fine wrinkles but no skin thickness; score 1="mild" skin thickness; score 2= "moderate" skin thickness with difficulty in making skin folds and no wrinkles; and score 3="severe" skin thickness with inability to make skin folds between 2 examining fingers. Where higher score indicating more severe disease.

SECONDARY OUTCOMES:
Change From Baseline in Forced Vital Capacity (FVC) at Week 52 | Baseline, at Week 52
  FVC will be assessed with the Flow screen spirometer.
Proportion of Responders to the Treatment Based on the Revised Composite Response Index in Systemic Sclerosis (rCRISS) at Week 52 | At Week 52
  Responders are defined as participants who meet all the following criteria: Improvement in 2 out of the 5 rCRISS components >=5% absolute increase from BL in ppFVC (percent predicted forced vital capacity), >=25% relative decrease from BL in mRSS, Health Assessment Questionnaire Disability Index (HAQ-DI), PGA (Patient's Global Assessment), CGA(Clinician/Physician's Global Assessment) score. Worsening in no more than 1 rCRISS component >=5% absolute decrease from BL in ppFVC, >=25% relative increase from BL in mRSS, HAQ-DI, PGA, CGA score. No significant SSc-related event.
Change From Baseline in mRSS at Weeks 8, 12, 24, 28, 36, 44, 52 | Baseline, at Week 8, 12, 24, 28, 36, 44, 52
  mRSS is the assessment of skin involvement includes semiquantitative estimation of skin thickness, pliability (hardness), and fixation to underlying structures (tethering).Cutaneous thickness is assessed in 17 body surface areas using a 0-3 scale, where mRSS of score 0="normal" with fine wrinkles but no skin thickness; score 1="mild" skin thickness; score 2= "moderate" skin thickness with difficulty in making skin folds and no wrinkles; and score 3="severe" skin thickness with inability to make skin folds between 2 examining fingers. Where higher score indicating more severe disease.
Percent change from Baseline in mRSS at Week 52 | Baseline, at Week 52
  mRSS is the assessment of skin involvement includes semiquantitative estimation of skin thickness, pliability (hardness), and fixation to underlying structures (tethering).Cutaneous thickness is assessed in 17 body surface areas using a 0-3 scale, where mRSS of score 0="normal" with fine wrinkles but no skin thickness; score 1="mild" skin thickness; score 2= "moderate" skin thickness with difficulty in making skin folds and no wrinkles; and score 3="severe" skin thickness with inability to make skin folds between 2 examining fingers. Where higher score indicating more severe disease.
Change from Baseline in Percent Predicted FVC (ppFVC) at Week 52 | Baseline, at Week 52
  FVC will be assessed with the Flow screen spirometer.
Percent Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 52 | Baseline, at Week 52
  HAQ-DI is a participant-reported questionnaire and sensitive to change in disease activity (cutaneous and visceral involvement and with changes in physiological parameters over time).Each question is rated on a 0 to 3 scale (0 = without difficulty; 3 = unable to do), and additional points can be added if aids or devices (i.e., cane, walker) are needed for specific activities. An increased score indicated worse functionality.
Percent Change From Baseline in Patient's Global Assessment (PGA) Score at Week 52 | Baseline, at Week 52
  The participant's global impression of health Numeric Rating Scale 0-10 (NRS) will be self-administered by the participant. 0 represents excellent and 10 represents extremely poor.
Percent Change From Baseline in Clinician's Global Assessment (CGA) Score at Week 52 | Baseline, at Week 52
  The clinician global impression of health Numeric Rating Scale 0-10 (NRS) will be filled out by the participant's clinician after all other study procedures have been completed. 0 represents excellent and 10 represents extremely poor.
Incidence and Severity of TEAEs, Treatment-Emergent SAEs, Treatment-Emergent AEs of Special Interest (AESIs), Significant SSc-Related TEAEs, TEAEs Leading to Investigational Product Discontinuation and Study Discontinuation. | From baseline of study intervention to 12 weeks after last dose (52 weeks)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A Serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: Results in death, life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect, Other serious (important medical events).
Incidence of Abnormal Vital Signs | From baseline of study intervention to 12 weeks after last dose (52 weeks)
  Change from BL in pulse rate, blood pressure, respiration rate, and body temperature will be assessed by visit and treatment group including participants with treatment emergent changes.
Incidence of Abnormal Laboratory Parameters | From baseline of study intervention to 12 weeks after last dose (52 weeks)
  Change from BL in hematology, clinical chemistry, and lipid variables will be assessed by visit and treatment group including participants with treatment-emergent changes.
Incidence of Abnormal Electrocardiogram (ECG) Findings | From baseline of study intervention to 12 weeks after last dose (52 weeks)
  Observed values of heart rate, QRS duration, PR interval, RR interval and QT interval will be summarized by visit and treatment group including participants with clinically significant abnormal results.
Incidence of Abnormal Weight Change | From baseline of study intervention to 12 weeks after last dose (52 weeks)
  Change from BL in weight (kilograms) will be assessed by visit and treatment and medically significant changes will be recorded as adverse events.

IPD SHARING:
Plan to Share IPD: No